CLINICAL TRIAL: NCT01901887
Title: The Better Resiliency Among Veterans With Omega-3's (BRAVO) Study: A Double Blind, Placebo-Controlled Trial of Omega-3 Fatty Acid Supplementation Among Military Veterans
Brief Title: The Better Resiliency Among Veterans With Omega-3's (BRAVO) Study
Acronym: BRAVO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Medical University of South Carolina (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bernadette Marriott, Professor Department of Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRAVO2013
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Suicide
Keywords: Adults; Suicidality
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Juice (Experimental): 3,300 mg of Omega-3 HUFAs per day for 6 months
  Other names: none
  Interventions: Drug: Study Juice
- Placebo Juice (Placebo Comparator): 3,300 mg of macadamia nut oil per day for 6 months
  Other names: none
  Interventions: Drug: Placebo Juice

INTERVENTIONS:
Drug: Study Juice — The intervention will be 3 boxes/day for 6 months of SMARTFISH® Nutrifriend 1100, a commercially available smoothie juice box containing 1,100 mg of omega-3 HUFAs/200 ml box (approximately 550 mg EPA and 550 mg DHA/box) for a total of 3,300 mg of omega-3 HUFAs/day (approximately 1,650 mg EPA and 1,650 mg DHA/day).
  Other Names: SMARTFISH® Nutrifriend 1100; Omega-3 formulated juice
  Arms: Study Juice
Drug: Placebo Juice — The placebo will be 3 boxes/day for 6 months of a placebo juice which will be identical to the study juice except that it will substitute 1,100 mg of macadamia nut oil/200 ml juice box in place of the omega-3 HUFAs for a total of 3,300 mg of macadamia nut oil/day.
  Other Names: Other names: Smartfish (placebo juice)
  Arms: Placebo Juice

SUMMARY:
The BRAVO study seeks to determine if dietary supplementation with omega-3 highly unsaturated fatty acids (omega-3 HUFAs) reduces the risk for serious suicidal behaviors, suicidal thinking, negative emotions, and symptoms associated with suicide risk, in a Veteran and non-Veteran population that is at risk for suicidal behaviors. This study seeks to evaluate the efficacy of omega-3 HUFAs among a representative population of US Veterans and non-Veterans already receiving appropriate medical care so that if successful, these results can be readily applied to broader populations in the US.

DETAILED DESCRIPTION:
The BRAVO study seeks to determine if dietary supplementation with omega-3 highly unsaturated fatty acids (omega-3 HUFAs) reduces the risk for serious suicidal behaviors, suicidal thinking, negative emotions, and symptoms associated with suicide risk, in a Veteran and non-Veteran population that is at risk for suicidal behaviors. Changes in cognitive processes specific to suicide risk will be evaluated, including implicit associations, response inhibition and sustained attention. Sub-analyses will evaluate efficacy in reducing depressive symptoms, alcohol and nicotine use among Veterans and non-Veterans with concomitant significant depressive symptoms, and alcohol and nicotine use disorders. In addition, a sub-study will utilize functional magnetic resonance imaging (fMRI) to evaluate the neuropsychological and neurophysiological effects of the omega-3 HUFAs. This study seeks to evaluate the efficacy of omega-3 HUFAs among a representative population of US Veterans and non-Veterans already receiving appropriate medical care so that if successful, these results can be readily applied to broader populations in the US.

ELIGIBILITY:
Inclusion criteria- Primary study

1. a Veteran or non-Veteran identified as being at risk for suicide and presently under the care of a mental healthcare provider (A release of information from his/her mental healthcare provider is required.)
2. age 18 - 90
3. within the participant's medical history, either

   1. a suicide attempt in the last 6 months, or
   2. a suicide attempt during the adult lifetime AND current diagnosis of an episode of depression as diagnosed on the Mini International Neuropsychiatric Interview (MINI), or
   3. an inpatient admission with suicide risk in the last 6 months, or
   4. an inpatient admission with suicide risk during the adult lifetime AND current diagnosis of an episode of depression as diagnosed on the Mini International Neuropsychiatric Interview (MINI), or
   5. positive suicidal behavior or ideation based on a psychiatrist- administered Columbia-Suicide Severity Rating Scale (C-SSRS) and psychiatrist review of participant medical history and physical], or
   6. a score of 0 or greater on the Implicit Associations Test-Suicide (IAT-S), or
   7. > or = 9 on the Beck Hopelessness Scale (BHS) and psychiatrist review of participant medical history and physical
4. participant can safely eat walnuts, pecans, almonds, peanuts and all other nuts
5. participant can safely eat apples, peaches, pears, pomegranates, aronia, jackfruit, and passion fruit
6. participant can safely eat the herb rosemary, and the fish salmon, trout and cod
7. participant can safely drink and eat food that contain whey and/or milk protein
8. willingness to drink the juice boxes 3 times each day for 6 months
9. have a stable residence with adequate space to store the juice
10. capacity to provide written informed consent

Additional inclusion criteria for Depressive Symptoms sub-analysis

1. enrollment in the primary study of suicide risk reduction
2. a Beck Depression Inventory ≥30
3. a diagnosis of a depressive disorder

Additional inclusion criteria for Alcohol and Nicotine use sub-analysis

1. enrollment in the primary study of suicide risk reduction
2. diagnosis of an alcohol use disorder or "at risk drinking patterns"
3. self-report of smoking >10 cigarettes/d.

Exclusion criteria-

1. unstable medical conditions requiring immediate attention or medical conditions that preclude potential study participation for the duration of the study
2. history of seizures, except for:

   * febrile seizures during childhood
   * history of a single seizure episode as an adult if not being maintained on anti-seizure medication; this single seizure must not be related to a primary seizure disorder (must not be epilepsy)
3. persons who have received a diagnosis of diabetes
4. those taking Isotretinoin (Accutane)
5. allergy, hypersensitivity, or intolerance to fish oils or omega-3 fats
6. allergy, hypersensitivity, or intolerance to Macadamia nuts or any nuts such as almonds, walnuts, pecans, peanuts, etc.
7. allergy, hypersensitivity, or intolerance to apples, peaches, pears, pomegranates, aronia, jackfruit, and passion fruit
8. allergy, hypersensitivity, or intolerance to the herb rosemary, and the fish: salmon, trout and cod
9. allergy, hypersensitivity, or intolerance to whey and/or milk protein
10. life threatening medical conditions or life expectancy of less than 6 months
11. pregnancy or lactation or intention to become pregnant within the next 12 months
12. acute intoxication or withdrawal from alcohol or other substances (to be determined by a clinical team member)
13. a cognitive impairment severe enough to preclude informed consent or valid responses on self-report questionnaires
14. Body Mass Index (BMI) <18 or >45
15. evidence of disordered eating or risk of malnutrition based on the Eating Attitudes Test (EAT-26)
16. relapsing of remitting Multiple Sclerosis
17. unstable or rapidly progressive neurological disease
18. history of significant behavioral instability
19. participating in another research study
20. regular use of anticoagulants such as high dose aspirin, warfarin or Coumadin
21. take hypoglycemic agents

Additional exclusion criteria for fMRI Study only (40 individuals)

* inability or unwillingness to participate in an fMRI scan
* presence of metallic objects in the body that would interfere with the scan
* pronounced claustrophobia
* body weight >300 pounds

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Impact of omega-3 HUFA supplementation on suicidal behaviors and thinking among adults. | 6 months
  Examine to see if dietary supplementation with omega-3 HUFAs results in fewer episodes of a New Episode of Significant Suicide Risk (NESSR)*, reduces symptom assessment scores for suicidality, reduces implicit associations with suicide and death, and improves performance scores on suicide related cognition tests.
  * A NESSR is defined as the occurrence of any of the following: a) a suicide death, or b) a suicide attempt, or c) an inpatient admission with suicide risk, or d) a "new VA medical record flag for suicidality", or outside the VA system a clinical diagnostic equivalent (the Columbia-Suicide Severity Rating Scale) and psychiatrist review of participant medical history and physical.

SECONDARY OUTCOMES:
Impact of omega-3 HUFA supplementation on symptoms of negative affect associated with suicide risk among adults. | 6 months
  Examine to see if dietary supplementation with omega-3 HUFAs reduces symptoms of perceptions of daily stress, anxiety, depression, and hopelessness.
Impact of omega-3 HUFA supplementation on symptoms of post-traumatic stress disorder (PTSD) associated with suicide risk among adults. | 6 months
  Examine to see if dietary supplementation with omega-3 HUFAs lowers the number of moderate to severe symptoms of PTSD, and decreases the severity of symptoms of PTSD among subjects with moderate to severe symptoms.
Impact of omega-3 HUFA supplementation on symptoms of cognitive functioning associated with suicide risk among adults. | 6 months
  Examine to see if dietary supplementation with omega-3 HUFAs improves sustained attention, response inhibition, and cognitive control; determine if changes in cognitive parameters are associated with changes in negative affect; and, determine if cognitive changes are associated with changes in suicide parameters.

OTHER OUTCOMES:
Impact of omega-3 HUFA supplementation among subjects with moderate to severe depressive symptoms to evaluate efficacy for clinically significant depressive symptoms. | 6 months
  Examine to see if higher blood levels of omega-3 HUFAs correlate with scores on the Beck Depression Inventory, and increase likelihood of a 50% reduction in depressive symptoms.
Impact of dietary supplementation with omega-3 fatty acids on alcohol consumption in suicidal adults with alcohol use disorders. | 6 months
  Examine to see if dietary supplementation with omega-3 HUFAs decreases alcohol use in alcohol-dependent individuals; decreases alcohol consumption in non-alcohol-dependent individuals who endorse risky alcohol use in the past 12 months; decreases obsessive and compulsive thoughts about alcohol; and, decreases use of cigarettes among persons who smoke >10 cigarettes/day. Examine to see if decreases in alcohol consumption are associated with decreases in negative affect and impulsivity; and, if they are associated with decreased suicidal ideation/behaviors.
Impact of an omega-3 HUFA intervention on prefrontal hypo activation to risky decision-making and recall of past suicidal events in suicide attempters, using functional Magnetic Resonance Imaging (fMRI). | 6 months
  Determine if dietary supplementation with omega-3 fatty acids increases activation of frontal brain regions associated with risky decision-making (e.g., orbitofrontal cortex); and those associated with suicide attempt recall (e.g., medial prefrontal cortex.)
Suicidal ideation and behavior at 6-months post treatment-initiation by fMRI. | 6 months
  Determine if increases in frontal activation to risky decision-making and recall of past suicidal events from baseline to 6-months post treatment-initiation are associated with less suicidal ideation and behavior at > 6-months post treatment-initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Marriott, PhD, Principal Investigator — Medical University of South Carolina; Joseph R Hibbeln, MD, Principal Investigator — LMBB, NIAAA, NIH
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Hibbeln JR. Fish consumption and major depression. Lancet. 1998 Apr 18;351(9110):1213. doi: 10.1016/S0140-6736(05)79168-6. No abstract available. PMID 9643729
- [Background] Hibbeln JR, Linnoila M, Umhau JC, Rawlings R, George DT, Salem N Jr. Essential fatty acids predict metabolites of serotonin and dopamine in cerebrospinal fluid among healthy control subjects, and early- and late-onset alcoholics. Biol Psychiatry. 1998 Aug 15;44(4):235-42. doi: 10.1016/s0006-3223(98)00141-3. PMID 9715354
- [Background] McNamara RK, Carlson SE. Role of omega-3 fatty acids in brain development and function: potential implications for the pathogenesis and prevention of psychopathology. Prostaglandins Leukot Essent Fatty Acids. 2006 Oct-Nov;75(4-5):329-49. doi: 10.1016/j.plefa.2006.07.010. Epub 2006 Sep 1. PMID 16949263
- [Background] Blasbalg TL, Hibbeln JR, Ramsden CE, Majchrzak SF, Rawlings RR. Changes in consumption of omega-3 and omega-6 fatty acids in the United States during the 20th century. Am J Clin Nutr. 2011 May;93(5):950-62. doi: 10.3945/ajcn.110.006643. Epub 2011 Mar 2. PMID 21367944
- [Background] Hibbeln JR. Depression, suicide and deficiencies of omega-3 essential fatty acids in modern diets. World Rev Nutr Diet. 2009;99:17-30. doi: 10.1159/000192992. Epub 2009 Jan 9. No abstract available. PMID 19136836
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617